CLINICAL TRIAL: NCT04397094
Title: Theracal Versus Formocresol Pulpotomy in Primary Molars
Brief Title: Theracal Pulpotomy in Primary Molars
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mariem Wassel, Assistant professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FDASU-Rec ID 101612
Record Dates: First submitted 2020-05-17; First posted 2020-05-21 (Actual); Results first posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Deep Caries
Keywords: Theracal; formocresol; pulpotomy
MeSH Terms: interventions — formocresol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Theracal LC (Experimental): Theracal LC was used as a medicament to cover root stumps of asymptomatic thirty primary molars with vital pulp exposures. Teeth were followed up clinically and radiographically for 12 months.
  Interventions: Drug: Theracal LC
- Formocresol (Active Comparator): Formocresol was used as a medicament to cover root stumps of asymptomatic thirty primary molars with vital pulp exposures. Teeth were followed up clinically and radiographically for 12 months.
  Interventions: Drug: Formocresol

INTERVENTIONS:
Drug: Theracal LC — pulpotomy
  Arms: Theracal LC
Drug: Formocresol — Pulpotomy
  Arms: Formocresol

SUMMARY:
Light cured silicate based cement (theracal LC) pulpotomy was compared to formocresol pulpotomy in primary molars.

DETAILED DESCRIPTION:
sixty primary molars were either treated with Theracal LC or formocresol pulpotomy. Teeth were followed up clinicaly and radiographically for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* healthy, cooperative children
* mandibular primary molars with vital pulp exposures

Exclusion Criteria:

* clinical or radiographic evidence of irreversible pulpitis
* physiological root resorption

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-03-17 (Actual); Study Completion 2019-03-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Theracal LC | Formocresol
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Formocresol: Formocresol (1/5 th concentration) was used as a medicament to cover root stumps of asymptomatic thirty primary molars with vital pulp exposures. Teeth were followed up clinically and radiographically for 12 months.
  Formocresol: Pulpotomy
- Total: Total of all reporting groups
Arm/Group | Theracal LC | Formocresol | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 30 | 60
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.71 (0.59) | 5.56 (0.71) | 5.61 (0.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 17 | 15 | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Egypt | 30 | 30 | 60
radiographic and clinical examinations [Number; unit: participants] | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Clinical Examination
Description: Number of participants with tooth mobility, restoration loss, gingival swelling/fistula, pain on percussion.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Theracal LC: Theracal LC was used as a medicament to cover root stumps of asymptomatic thirty primary molars with vital pulp exposures. Teeth were followed up clinically and radiographically for 12 months.
  Theracal LC: pulpotomy
  NO clinical failures was evident over the 12 months follow up
- Formocresol: Formocresol was used as a medicament to cover root stumps of asymptomatic thirty primary molars with vital pulp exposures. Teeth were followed up clinically and radiographically for 12 months.
  Formocresol: Pulpotomy
  NO clinical failures was evident over the 12 months follow up
Arm/Group | Theracal LC | Formocresol
Number analyzed (Participants) | 30 | 30
Participants | 30 | 30

2. Secondary Outcome: Radiographic Examination
Description: Number of participants showing teeth with inter-radicular bone resorption, periapical bone resorption, internal root resorption, external root resorption, widening of periodontal ligament space.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Theracal LC | Formocresol
Number analyzed (Participants) | 30 | 30
Participants | 30 | 30

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Theracal LC | Formocresol
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 3/30 | 5/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Theracal LC (N=30) | Formocresol (N=30)
internal resorption (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
interradicular bone resorption (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-21): https://cdn.clinicaltrials.gov/large-docs/94/NCT04397094/Prot_SAP_000.pdf